CLINICAL TRIAL: NCT00612326
Title: Feasibility Evaluation of Magnetic Resonance Imaging and Positron Emission Tomography for Bladder Cancer Diagnosis and Staging
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03-024
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Bladder Cancer; Transitional Cell Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients with newly diagnosed locally or regionally advanced transitional cell carcinoma of the bladder.
  Interventions: Procedure: MRI and PET scanning procedures

INTERVENTIONS:
Procedure: MRI and PET scanning procedures — a CT scan, MRI, and C-11 Acetate PET scan. All these scans will be done as an outpatient. After you finish these scans, your doctor will schedule you for surgery to remove your bladder and lymph nodes.

SUMMARY:
The purpose of this study is to to find out if the MRI and PET scans can truly stage patients with bladder cancer. Both scans use newer ways to find out if your disease has grown beyond the bladder. The radioactive tracer used for the PET scan is called C-11 Acetate. We want to see if PET scan will be able to take a picture of the inside of your body that is better than other scans such as the CT scan and MRI. Therefore, the findings of the PET scan will be compared with other imaging studies as well as the surgical findings.

ELIGIBILITY:
Inclusion Criteria:

* Thirty (30) patients will be enrolled in this pilot study.
* All patients will have a clinical or histologic diagnosis of bladder cancer with active disease identified within the bladder at the time of consent and imaging.
* Patients with primary resectable lesions, and localized or regionally extensive disease will be eligible with residual disease in the bladder at the time of imaging.
* All patients will have consented to treatment at MSKCC

Exclusion Criteria:

* Prior pelvic radiation for bladder cancer
* Non-transitional cell histologies
* Patients deemed not appropriate surgical candidates
* Patients that are pregnant or lactating
* Patients that cannot tolerate being in the PET or MRI scanner for the duration of the study. Patients deemed unable to receive a contrast enhance CT will remain eligible.
* Vulnerable patients (minors, mentally retarded, prisoners, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited through the outpatient clinics of the Departments of Urology and Medical Oncology of MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2004-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the logistical and technical parameters that are needed to use 11C acetate-PET, and MRI for the preoperative detection of nodal metastases in patients with invasive bladder cancer. | conclusion of the study

SECONDARY OUTCOMES:
Evaluate the logistical and technical parameters needed to use contemporary pelvic MRI for preop primary tumor staging in pts with invasive disease (>T2) through detailed comparison of MRI imaging and pathologic findings following radical cystectomy. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Bochner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org